CLINICAL TRIAL: NCT05821335
Title: The Development and Investigation of Effectiveness of Leap Motion Based Gamefication Exercises in Hand Rehabilitation of the Individuals With Systemic Sclerosis
Brief Title: Leap Motion Based Gamefication Exercises in the Individuals With Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tugba Civi Karaaslan, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulC3
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Rheumatology; Scleroderma, Systemic; Video Games; Physiotherapy; Rehabilitation; Hand Rheumatism
Keywords: Scleroderma, Systemic; Hand therapy; Therapy, Computer-Assisted
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessment and treatment will be done by different investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leap motion assisted rehabilitation (Experimental): Individuals who will participate in the study will be treated 2 days a week for 5 weeks with Leap Motion sensor-supported games aimed at increasing patient-specific wrist flexion, wrist extension, ulnar and radial deviation of the wrist, flexion, extension and abduction of the fingers. Each training period will last 30 minutes.
  Interventions: Other: Leap motion assisted rehabilitation
- Traditional program (Experimental): They will be included in traditional rehabilitation training consisting of stretching exercises, strengthening exercises and functional exercises including activities of daily living for 2 days a week for 5 weeks.
  Interventions: Other: Traditional program

INTERVENTIONS:
Other: Leap motion assisted rehabilitation — Hand Therapy via leap motion sensor
  Arms: Leap motion assisted rehabilitation
Other: Traditional program — Hand Therapy by physiotherapist via traditional methods
  Arms: Traditional program

SUMMARY:
Leap Motion Based Gamefication Exercises in the Individuals With Systemic Sclerosis

DETAILED DESCRIPTION:
The aim of this project is to develop Leap Motion Sensor-assisted rehabilitation games that can be easily applied in hand rehabilitation in individuals with SSc, motivating, directing to the right exercise, providing therapeutic evaluation and feedback during the game, and comparing the effectiveness of these rehabilitation games with traditional rehabilitation applications.

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to adapt to exercises
* Not having any diagnosed cardiac or orthopedic disease that may prevent the application of assessment methods

Exclusion Criteria:

* Having a diagnosis of juvenile-onset SSc
* Having a history of neurological disease or trauma that will affect hand functions
* Receiving another treatment, such as intra-articular injection, surgery, that may affect hand rehabilitation in the last 6 months
* Having systemic involvement that may affect the treatment process or activities of daily living

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
modified Hand Mobility in Scleroderma (mHAMIS) | change from baseline at 5 weeks
  Hand Mobility in Scleroderma is a hand function test developed for adults who have systemic sclerosis. HAMIS consists of 9 items designed to measure all movements assessed in an ordinary range of motion-measured hand test. Each item is graded on a 0-3 scale, where 0 corresponds to normal function and 3 denotes that the individual is unable to perform the item. Each hand is assessed separately. The total score of HAMIS for each hand is 370 Sandqvist and Eklund Vol. 13, No. 6, December 2000 27, which represents a high degree of dysfunction.

SECONDARY OUTCOMES:
Finger Joint Range of Motion | change from baseline at 5 weeks
  The patients will be asked to close their fingers tightly and the distance between the pulp of the 2nd, 3rd, 4th, and 5th finger - distal palmar line (PP-DPD) will be measured in cm with the help of a ruler. Dominant and nondominant hand total scores will be calculated by summing the values found for the fingers of each hand separately.
Grip Strength | change from baseline at 5 weeks
  A hand dynamometer will be used. For measurements, patients will be asked to make a maximally voluntary grip while sitting, elbow flexed to 90 degrees, wrist in semi-pronation with thumb pointing up. Measurements on the sick and healthy hand will be made 3 times in a row, and the average values will be recorded in kilograms (kg). Finger grip will be evaluated with a pinchmeter in three different positions (lateral, palmar, fingertip).
Skin Hardness | change from baseline at 5 weeks
  Skin hardness will be measured with a durometer. Although the durometer is a device designed to measure non-biomaterial surface hardness, it is used clinically to evaluate sclerosis. Measurements will be made on the dorsal surface of the third finger, midphalanx, dorsum of the hand, palmar and dorsal aspects of the forearm.
Purdue Pegboard Test | change from baseline at 5 weeks
  Purdue Pegboard Test will be used to evaluate hand functions. This test is an objective and standardized test that is frequently used in practice to evaluate functional hand use. The test will be preferred because of its advantages in demonstrating the functional activities and ability of the hand and its ease of use. The patient will be asked to perform the test activities first with the dominant hand, then with the non-dominant hand in 30 seconds, and using both hands in 60 seconds. Scoring will be based on the number of successfully placed pins.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA CIVI KARAASLAN, PhD, Principal Investigator — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tarakci E, Arman N, Tarakci D, Kasapcopur O. Leap Motion Controller-based training for upper extremity rehabilitation in children and adolescents with physical disabilities: A randomized controlled trial. J Hand Ther. 2020 Apr-Jun;33(2):220-228.e1. doi: 10.1016/j.jht.2019.03.012. Epub 2019 Apr 19. PMID 31010703
- [Background] Murphy SL, Poole JL, Chen YT, Lescoat A, Khanna D. Rehabilitation Interventions in Systemic Sclerosis: A Systematic Review and Future Directions. Arthritis Care Res (Hoboken). 2022 Jan;74(1):59-69. doi: 10.1002/acr.24737. Epub 2021 Dec 22. PMID 34165263